CLINICAL TRIAL: NCT05510817
Title: Multiparametric Clinical, Radiological, Neuropsychological, and Neurophysiological Assessment to Investigate Prognostic Factors for Disease Evolution and Treatment Response in MS: a Prospective Study.
Brief Title: Multiparametric Assessment to Investigate Prognostic Factors for Disease Evolution a nd Evolutionary Patterns of Cognitive Status in RRMS
Acronym: COGNIT-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: Saint-Luc University Hospital (Unknown)
Responsible Party: Principal Investigator, Frédéric London, Principal Investigator, University Hospital of Mont-Godinne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B039202042775
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: MRI; evoked potentials; cognitive function; PROMs
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RRMS patients (Other): RRMS patients initiating a new DMT
  Interventions: Other: Multiparametric assessment

INTERVENTIONS:
Other: Multiparametric assessment — neuropsychological assessment, PRO measures, non-conventional MRI metrics

SUMMARY:
This prospective study combining non conventional MRI techniques, neuropsychological screening tools, and a neurophysiological work-up using a sensitive and validated battery, will evaluate the predictive value of these measures and will explore the changes of the cognitive scores from baseline.

DETAILED DESCRIPTION:
Neurologists are in need for reliable and robust predictive factors enabling to predict disease evolution and treatment response. Moreover, recent studies suggested that the evolution patterns of cognitive status in MS could be mixed, contradicting the concept that cognitive impairment in MS will inevitably increase over time.

The main aim of this prospective study is to investigate the predictors of disease evolution, as measured by the EDSS score, using a multiparametric assessment combining neuropsychological tests (BCcogSEP battery), MRI-derived metrics (volumetric brain parameters, tractography, diffusion tensor imaging and fiber tracking), patient-reported outcome measures, and neurophysiological tools (multimodal evoked potentials), and to explore the evolutionary patterns of cognitive status (changes from baseline).

The investigators planned to include 50 patients with active RRMS and initiating a new disease-modifying treatment.

Yearly assessment starting from study inclusion will be performed.

ELIGIBILITY:
Inclusion Criteria:

* active MS, according to the Lublin criteria
* disease duration < 10 years before initiating or changing a disease-modifying therapies,
* relapse- and steroid-free for at least 1 month before MRI acquisition
* between 18-50 years old
* having given informed consent
* with no significant comorbidity other than MS or substance abuse that could interfere with cognitive performances

Exclusion Criteria:

* progressive forms of MS

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Predictors of disease evolution | 3 years
  EDSS score worsening from baseline
evaluation of evolutionary patterns of cognitive status (impaired vs non impaired)/changes from baseline | 3 years
  changes from baseline in cognitive scores
baseline predictors of future cognitive impairment | 3 years
  abnormal cognitive performances based on cognitive scores (using BCcogSEP battery)

SECONDARY OUTCOMES:
alteration in strategic white matter tracts at the early stages of RRMS, in patients with and without cognitive impairment | 3 years
  fractional anisotropy
predictive role of mEPS in predicting future disability | 3 years
  the Global Evoked Potential (GEP) score at study entry (baseline); EDSS score changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric London, MD, Principal Investigator — University Hospital Mont-Godinne
Locations (1):
- CHU UCL Namur site Godinne, Yvoir, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No